CLINICAL TRIAL: NCT01104779
Title: A Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of Cariprazine in the Acute Exacerbation of Schizophrenia
Brief Title: Safety and Efficacy of Cariprazine in Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGH-MD-05
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Acute Schizophrenia; Psychotropic Drugs; Antipsychotic Agents; Mental Disorders; Dopamine Agents; Central Nervous System Agents
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cariprazine (3-6 mg/day) (Experimental): Cariprazine once daily fixed-flexible low dose
  Interventions: Drug: Cariprazine
- Cariprazine (6-9 mg/day) (Experimental): Cariprazine once daily fixed-flexible high dose
  Interventions: Drug: Cariprazine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Patients who meet eligibility criteria will be administered a once daily oral dose of cariprazine for six weeks. Upon completion of the study or early termination, patients will undergo a two week safety follow-up period.
  Other Names: RGH-188
  Arms: Cariprazine (3-6 mg/day); Cariprazine (6-9 mg/day)
Drug: Placebo — Patients who meet eligibility criteria will be administered a once daily oral dose of placebo for six weeks. Upon completion of the study or early termination, patients will undergo a two week safety follow-up period.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, and tolerability of cariprazine relative to placebo for the treatment of acute exacerbation of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided informed consent prior to any study specific procedures
* Patients currently meeting the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for schizophrenia (paranoid type, disorganized type, catatonic type or undifferentiated type), as confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (SCID)
* Structured Clinical Interview for the Positive and Negative Syndrome Scale (SCIPANSS) total score ≥ 80 and ≤ 120
* Diagnosis of schizophrenia for a minimum of 1 year before Visit 1
* Patients with normal physical examination, laboratory, vital signs,and/ or electrocardiogram (ECG)

Exclusion Criteria:

* Patients with a DSM-IV-TR diagnosis of Schizoaffective disorder, schizophreniform disorder, other psychotic disorders other than schizophrenia, or bipolar I or II disorder
* Patients in their first episode of psychosis
* Pregnant, breast-feeding, and/or planning to become pregnant and/or breastfeed during the study
* Pervasive developmental disorder, mental retardation, delirium, dementia, amnestic and other cognitive disorders
* Known or suspected borderline or antisocial personality disorder or other DSM-IV-TR axis II disorder of sufficient severity to interfere with participation in this study
* Substance abuse or dependence within the prior 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 446 (Actual)
Dates: Start 2010-04-27 (Actual); Primary Completion 2011-12-15 (Actual); Study Completion 2011-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Migliore, MA, Study Director — Forest Laboratories
Locations (41):
- United States (15):
  - Forest Investigative Site 48, Costa Mesa, California
  - Forest Investigative Site 50, Long Beach, California
  - Forest Investigative Site 42, Paramount, California
  - Forest Investigative Site 054, San Diego, California
  - Forest Investigative Site 41, Kissimmee, Florida
  - Forest Investigative Site 055, Atlanta, Georgia
  - Forest Investigative Site 44, Rockville, Maryland
  - Forest Investigative Site 45, St Louis, Missouri
  - Forest Investigative Site 52, Las Vegas, Nevada
  - Forest Investigative Site 40, Cedarhurst, New York
  - Forest Investigative Site 46, Cincinnati, Ohio
  - Forest Investigative Site 47, Philadelphia, Pennsylvania
  - Forest Investigative 49, Memphis, Tennessee
  - Forest Investigative Site 51, Houston, Texas
  - Forest Investigative Site 43, Irving, Texas
- Colombia (4):
  - Forest Investigative Site 601, Bello, Antioquia
  - Forest Investigative Site 604, Pereira, Risaralda Department
  - Forest Investigative Site 602, Bogotá
  - Forest Investigative Site 605, Bogotá
- India (19):
  - Forest Investigative Site 505, Vijayawada, Andhra Pradesh
  - Forest Investigative Site 514, Visakhapatnam, Andhra Pradesh
  - Forest Investigative Site 503, Ahmedabad, Gujarat
  - Forest Investigative Site 519, Ahmedabad, Gujarat
  - Forest Investigative Site 501, Ahmedabad, Gujarat
  - Forest Investigative Site 508, Ahmedabad, Gujarat
  - Forest Investigative Site 504, Bangalore, Karna
  - Forest Investigative Site 517, Mangalore, Karna
  - Forest Investigative Site 515, Mangalore, Karna
  - Forest Investigative Site 516, Mysore, Karna
  - Forest Investigative Site 500, Aurangabad, Mahara
  - Forest Investigative Site 510, Mumbai, Mahara
  - Forest Investigative Site 513, Nashik, Mahara
  - Forest Investigative Site 511, Pune, Mahara
  - Forest Investigative Site 502, Pune, Mahara
  - Forest Investigative Site 509, Rajkot, Rajasthan
  - Forest Investigative Site 507, Kanpur, Uttar Pradesh
  - Forest Investigative Site 518, Lucknow, Uttar Pradesh
  - Forest Investigative Site 506, Varanasi, Uttar Pradesh
- South Africa (3):
  - Forest Investigative Site 704, Johannesburg, Gauteng
  - Forest Investigative Site 703, Cape Town, W Cape
  - Forest Investigative Site 706, Cape Town, W Cape

REFERENCES:
- [Derived] Laszlovszky I, Barabassy A, Nemeth G. Cariprazine, A Broad-Spectrum Antipsychotic for the Treatment of Schizophrenia: Pharmacology, Efficacy, and Safety. Adv Ther. 2021 Jul;38(7):3652-3673. doi: 10.1007/s12325-021-01797-5. Epub 2021 Jun 6. PMID 34091867
- [Derived] Barabassy A, Sebe B, Acsai K, Laszlovszky I, Szatmari B, Earley WR, Nemeth G. Safety and Tolerability of Cariprazine in Patients with Schizophrenia: A Pooled Analysis of Eight Phase II/III Studies. Neuropsychiatr Dis Treat. 2021 Apr 7;17:957-970. doi: 10.2147/NDT.S301225. eCollection 2021. PMID 33854317
- [Derived] Marder S, Fleischhacker WW, Earley W, Lu K, Zhong Y, Nemeth G, Laszlovszky I, Szalai E, Durgam S. Efficacy of cariprazine across symptom domains in patients with acute exacerbation of schizophrenia: Pooled analyses from 3 phase II/III studies. Eur Neuropsychopharmacol. 2019 Jan;29(1):127-136. doi: 10.1016/j.euroneuro.2018.10.008. Epub 2018 Nov 20. PMID 30470662
- [Derived] Earley W, Durgam S, Lu K, Laszlovszky I, Debelle M, Kane JM. Safety and tolerability of cariprazine in patients with acute exacerbation of schizophrenia: a pooled analysis of four phase II/III randomized, double-blind, placebo-controlled studies. Int Clin Psychopharmacol. 2017 Nov;32(6):319-328. doi: 10.1097/YIC.0000000000000187. PMID 28692485
- [Derived] Cutler AJ, Durgam S, Wang Y, Migliore R, Lu K, Laszlovszky I, Nemeth G. Evaluation of the long-term safety and tolerability of cariprazine in patients with schizophrenia: results from a 1-year open-label study. CNS Spectr. 2018 Feb;23(1):39-50. doi: 10.1017/S1092852917000220. Epub 2017 May 8. PMID 28478771
- [Derived] Citrome L, Durgam S, Lu K, Ferguson P, Laszlovszky I. The effect of cariprazine on hostility associated with schizophrenia: post hoc analyses from 3 randomized controlled trials. J Clin Psychiatry. 2016 Jan;77(1):109-15. doi: 10.4088/JCP.15m10192. PMID 26845266

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization and treatment assignment were based on a randomization scheme prepared by Allergan Biostatistics prior to the start of the study. No-drug washout period of up to 7 days.
Groups:
- Placebo; Cariprazine (3-6 mg/Day); Cariprazine (6-9 mg/Day): Oral administration. Once per day.
Period: Overall Study
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-9 mg/Day)
Started | 147 | 151 | 148
Completed | 88 | 96 | 86
Not Completed | 59 | 55 | 62
Not completed — Protocol Violation | 1 | 2 | 2
Not completed — Lack of Efficacy | 26 | 12 | 13
Not completed — Adverse Event | 13 | 14 | 13
Not completed — Did not meet inc/exc criteria | 1 | 1 | 1
Not completed — Other reasons | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Withdrawal by Subject | 16 | 25 | 32

BASELINE CHARACTERISTICS:
Population: The randomized population is also the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-9 mg/Day) | Total
Number analyzed (Participants) | 147 | 151 | 148 | 446
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.7 (11.3) | 36.6 (10.5) | 35.5 (9.3) | 36.3 (10.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 110 | 118 | 113 | 341
  Female | 37 | 33 | 35 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 24 | 27 | 74
  Not Hispanic or Latino | 124 | 127 | 121 | 372
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 28 | 30 | 84
  Black or African-American | 51 | 56 | 53 | 160
  Asian | 56 | 56 | 56 | 168
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 3
  Other | 12 | 10 | 6 | 28

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Schizophrenia Symptoms: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The Positive and Negative Syndrome Scale is a 30-item rating scale specifically developed to asses both the positive and negative symptom syndromes of patients with schizophrenia. The PANSS total score is rated based on a structured clinical interview with the patient and supporting clinical information obtained from family, hospital staff, or other reliable informants. This assessment provides scores in 9 clinical domains, including a positive syndrome, a negative syndrome, depression, a composite index, and general psychopathology. Each item is scored on a 7-point (1 to 7) scale, with 1 being minimal impact, and 7 being highest impact. The cumulative score ranges from 30 to 210. A negative change score indicates improvement.
Time Frame: Baseline to Week 6
Population: Intent-to-Treat Population, consisting of all patients in the Safety Population who had at least one postbaseline assessment of the PANSS total score.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-9 mg/Day)
Number analyzed (Participants) | 145 | 147 | 147
Units on a Scale | -16.0 (1.6) | -22.8 (1.6) | -25.9 (1.7)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine (3-6 mg/Day); Test type: Superiority; p = 0.0029, ANCOVA; Mean Difference (Final Values) = -6.8, 95% CI 2-sided [-11.3 to -2.4] — Cariprazine 3-6 mg/day vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Cariprazine (6-9 mg/Day); Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -9.9, 95% CI 2-sided [-14.5 to -5.3] — Cariprazine 6-9 mg/day vs Placebo

2. Secondary Outcome: Measurement of Schizophrenia Symptoms: Change From Baseline in Clinical Global Impression-Severity (CGI-S)
Description: The Clinical Global Impressions-Severity scale is a clinician-rated scale that measures the overall severity of a participant's illness in comparison with the severity of illness in other participants the physician has observed. The participant is rated on a scale from 1 to 7 with 1 indicating a "normal state" and 7 indicating "among the most extremely ill participants." A higher score indicates greater illness. A negative change score indicates improvement.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-9 mg/Day)
Number analyzed (Participants) | 145 | 147 | 147
units on a scale | -1.0 (0.1) | -1.4 (0.1) | -1.6 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine (3-6 mg/Day); Test type: Superiority; p = 0.0115, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to -0.1] — Cariprazine 3-6 mg/day vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Cariprazine (6-9 mg/Day); Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.8 to -0.3] — Cariprazine 6-9 mg/day vs Placebo

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for 8 weeks.
Description: Safety Population: All patients in the randomized population who took at least 1 dose of double-blind investigational product.
Arm/Group | Placebo | Cariprazine (3-6 mg/Day) | Cariprazine (6-9 mg/Day)
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/151 | 0/148
Serious Adverse Events (participants affected / at risk) | 13/161 | 9/167 | 4/169
Other Adverse Events (participants affected / at risk) | 54/147 | 84/151 | 86/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | Cariprazine (3-6 mg/Day) (N=167) | Cariprazine (6-9 mg/Day) (N=169)
Psychotic disorder (Psychiatric disorders) | 2 | 4 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 3 | 3 | 0
Schizophrenia (Psychiatric disorders) | 6 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Polydipsia psychogenic (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | Cariprazine (3-6 mg/Day) (N=151) | Cariprazine (6-9 mg/Day) (N=148)
Nausea (Gastrointestinal disorders) | 7 | 7 | 14
Constipation (Gastrointestinal disorders) | 5 | 14 | 10
Dyspepsia (Gastrointestinal disorders) | 6 | 3 | 10
Vomiting (Gastrointestinal disorders) | 4 | 8 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 8 | 6
Weight increased (Investigations) | 2 | 5 | 8
Akathisia (Nervous system disorders) | 5 | 24 | 25
Headache (Nervous system disorders) | 19 | 14 | 24
Extrapyramidal disorder (Nervous system disorders) | 4 | 8 | 15
Tremor (Nervous system disorders) | 3 | 12 | 8
Insomnia (Psychiatric disorders) | 16 | 10 | 16
Restlessness (Psychiatric disorders) | 7 | 10 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.